CLINICAL TRIAL: NCT01987323
Title: Safety and Efficacy of Liposomal Latanoprost in Ocular Hypertensive Patients
Brief Title: Safety and Efficacy of Liposomal Latanoprost in Ocular Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Principal Investigator, A/Prof Tina Wong, Associate Professor, Singapore Eye Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R967/76/2012
Record Dates: First submitted 2013-10-30; First posted 2013-11-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Ocular Hypertension
Keywords: glaucoma; raised intraocular pressure
MeSH Terms: conditions — Ocular Hypertension; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lipolat (Experimental): Subconjunctival injection of Lipolat into the superior bulbar conjunctiva of all enrolled participants
  Interventions: Drug: Subconjunctival injection of liposomal latanoprost

INTERVENTIONS:
Drug: Subconjunctival injection of liposomal latanoprost

SUMMARY:
Aim: Evaluation of a single subconjunctival injection of liposomal EggPC formulation of latanoprost in treating glaucoma.

Hypothesis: The investigators have already evaluated carrier stability, drug partitioning, in vitro drug release, tolerance, and efficacy of latanoprost-incorporated EggPC liposomes upon subconjunctival administration in both rabbit and monkey eyes. Therefore, the investigators hypothesize that this would be safe and efficacious in humans as well.

Methodology: A pilot study to assess a liposome formulation containing latanoprost. The investigators will recruit 6 study subjects with eyes that have raised IOP, for subconjunctival injection of this liposome formulation. The recruited eye will be injected and monitored for inflammation, toxicity and pain as primary end-points. Monitoring of the eye will be for the first 24 hours post-injection, week 2, months 1, 2 and 3 thereafter.

Importance: If proven safe, this method of drug delivery could potentially be used for treatment of raised intraocular pressures in blinding conditions such as glaucoma.

DETAILED DESCRIPTION:
The number of recorded adverse events and intolerance to the subconjunctival injection procedure by the participants during the study period was used as a measure of safety.

ELIGIBILITY:
Inclusion Criteria:

Glaucoma patients who have eyes with raised IOP (baseline IOP >21 mmHg) due to end-stage glaucoma with a poor visual prognosis.

Exclusion criteria:

1. Active or recent eye infection, endophthalmitis
2. Known hypersensitivity to latanoprost
3. Only eye
4. Previous glaucoma filtration surgeries or trabeculectomy
5. Intraocular pressure less than 12mmHg.
6. Inability to give informed consent.
7. Inability to safely administer a subconjunctival injection
8. Uncontrolled systemic hypertension, CVA or TIA within the previous month.
9. Pregnancy -

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious adverse events | 3 months

SECONDARY OUTCOMES:
intraocular pressure | 3 months
  Intraocular pressure reduction from baseline pressure reading

CONTACTS AND LOCATIONS:
Overall Officials: Tina T Wong, MD, PhD, Principal Investigator — Singapore National Eye Centre

REFERENCES:
- See also: Related Info — https://eservice.hsa.gov.sg/prism/ct_r/enquiry.do?action=getAllTherapeuticArea